CLINICAL TRIAL: NCT02825173
Title: A Prospective, Multi-center, Open Label, Non-randomized Study, of Seal-G Surgical Sealant for the Reinforcement of Gastrointestinal Anastomosis
Brief Title: Seal-G Safety Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sealantis Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DLG-072-01
Record Dates: First submitted 2016-06-15; First posted 2016-07-07 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Elective Surgical Procedures, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Seal-G (Experimental): A surgical sealant intended for use as an adjunct to standard closure techniques for reinforcement and protection of gastrointestinal anastomoses.
  Interventions: Device: Seal-G

INTERVENTIONS:
Device: Seal-G — Intervention:
  Device: Seal-G Seal-G is applied adjunctively to cover standard closure techniques
  Other Names: Seal-G Surgical Sealant

SUMMARY:
The purpose of this study is to farther assess the safety of the Seal-G Surgical Sealant for the reinforcement and protection of gastrointestinal anastomosis.

DETAILED DESCRIPTION:
Pre-Surgery:

Screening will be performed among adult subjects who are scheduled for an elective colorectal surgery. Pre-surgery assessments (after completion of consent process and signed ICF) will be according to the routine practice.

Intra-operative:

During surgery, an assessment of the intra-operative exclusion criteria will be performed. If the subject does not meet any of the exclusion criteria, the subject will be further enrolled. Surgery will be performed according to the site standard of care (routine practice). Anastomosis will be created either using a stapler device (linear or circular), according to manufacture IFU (Instructions for use) or hand suture according to surgeon best practice technique. Once anastomosis has been created, surgeon will verify the anastomosis and mucosal donuts integrity.

Device (Seal-G) application on anastomotic site

Post-operative follow-up: Follow-up evaluations will be performed daily while hospitalized. There will be one postoperative follow up at one month - clinic visit

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old.
2. Subject is planned to undergo an elective open or laparoscopic colonic resection with the creation of an anastomosis (extracorporeal if laparoscopic surgery is performed).
3. Subject signs and dates a written ICF, indicates an understanding of the study procedures and follow-up requirements and is willing to comply with them.

Exclusion Criteria:

1. Subject, undergoing low anterior resection
2. Subject is planned to undergo an emergency procedure
3. Subject has a diagnosis of bowel strangulation, peritonitis, bowel perforation, local or systemic infection, ischemic bowel, and carcinomatosis
4. Subject treated with immunosuppressive agents within 28 days prior to study enrollment (including corticosteroids)
5. Serious or uncontrolled co-existent diseases (e.g. severe cardiovascular disease, congestive heart failure, recent myocardial infarction, significant vascular disease, active or uncontrolled autoimmune disease, active or uncontrolled infection)
6. Subject who according to the investigator clinical judgement is at risk for anastomosis dehiscence
7. Subject has participated in another clinical study which may affect this study's outcomes within the last 30 days
8. Subject's ASA (American Society of Anesthesiology) score ≥ 4
9. Subject's BMI > 34 or <16
10. Subject known to have distant metastases, such as liver, lung, bone etc. metastases (not including local and regional lymph nodes)
11. Subject with a life expectancy of less than 1 year
12. Subject requires more than one anastomosis during the surgery
13. Woman who is known to be pregnant
14. Mentally handicapped, prisoners, or legally incompetent

Intraoperative Exclusion Criteria:

1. Subjects whom anastomosis is less than 10 cm from the anal verge
2. The full circumference of the anastomosis is not accessible for Seal-G application
3. Subject received intraoperative sealant, glue or any buttressing material for the study related anastomosis, other than the Seal-G
4. Subject has excessive intraoperative bleeding prior to the anastomosis formation as assessed by the investigator (estimated in excess of 500mL)
5. Subject has peritoneal carcinomatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08; Primary Completion 2016-11 (Actual); Study Completion 2016-12-02 (Actual)

PRIMARY OUTCOMES:
Rate of device related complications | Postoperative to end of follow up (30±7 days)

SECONDARY OUTCOMES:
Overall rate of complications | Postoperative to end of follow up (30±7 days)
Postoperative length of hospitalization stay | Postoperative till time for "ready to be discharged" (10±4 days)
Duration of sealant application | Intraoperative: starting from initial spreading on the treatment site to completion of curing, will be recorded (in minutes)
Ease of use of the device | Intraoperative: device application
  Ease of use of the device will be rated using a Likert scale from 1 to 5 with: 1 being Very easy, 2 Easy, 3 Neutral, 4 Difficult and 5 being Very difficult. At the day of surgery (after surgery completed) the surgeon will complete a questionnaire regarding the device use and ease of application.

CONTACTS AND LOCATIONS:
Overall Officials: Rina Lev, PhD, Study Director — Sealantis Ltd.
Locations (3):
- Israel (2):
  - Rabin Medical Center, Petah Tikva
  - Assaf Harofeh, Tzrifin
- Humanitas Research Hospital, Rozzano Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided